CLINICAL TRIAL: NCT03808467
Title: Transdiagnostic Cognitive Remediation Therapy for Patients With Eating Disorders: a Randomized Controlled Trial
Brief Title: Cognitive Training for Patients With Eating Disorders
Acronym: TCRTRCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/1182
Record Dates: First submitted 2018-12-18; First posted 2019-01-17 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder
Keywords: Cognitive Remediation; Neuropsychology; Neuropsychological Tests
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRT + TAU (Experimental): Cognitive Remediation Therapy + Treatment As Usual
  Interventions: Behavioral: Cognitive Remediation Therapy; Other: Treatment as usual
- TAU only (Other): Treatment As Usual
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy — Nine individual transdiagnostic CRT sessions will be delivered once per week, each session lasting approximately 45 minutes. Building on previously published CRT manuals for anorexia nervosa and obesity, a transdiagnostic CRT manual developed for this project will be used during the course of CRT treatment. The manual comprises an introduction to CRT for eating disorders, and a detailed nine-session structure incorporating cognitive and behavioral tasks in the following domains; (1) planning-impulsivity, (2) flexibility-rigidity and (3) central coherence-attention to details. A certain set of guiding questions will accompany each task with the aim of stimulating metacognition (i.e. thinking about thinking).
  Other Names: CRT
  Arms: CRT + TAU
Other: Treatment as usual — According to Norwegian guidelines established by the Norwegian Directorate of Health, the patients are likely to receive treatment focusing directly on the ED symptomatology, i.e normalization of weight in the case of underweight, reduction of binging and purging and normalization of other ED related thoughts and behaviors. Since both in-patients, patients in day treatment and out-patients will be included in the study, the number of hours with therapeutic interventions will vary. Records of the participants' received number of therapeutic hours will be logged weekly during the intervention for participants in both arms of the study.
  Other Names: TAU

SUMMARY:
Eating disorders are severe mental illnesses, mainly affecting adolescent- and young adult women. The prognoses for eating disorders are relatively poor, and a large part of patients with these illnesses do not benefit from available conventional therapies. After decades of research into the causes of eating disorders, there is now compelling evidence for specific neuropsychological difficulties in patients affected by eating disorders. These neuropsychological difficulties are characterized by cognitive and behavioral rigidity (poor set-shifting abilities), as well as difficulties related to central coherence, planning and impulse control. Surprisingly, few therapies specifically target these difficulties, and they are rarely incorporated into treatment. Cognitive Remediation Therapy has shown promising results as an adjunctive therapeutic intervention for patients with anorexia Nervosa. The primary aim of this randomized controlled trial is thus to investigate the effect of Cognitive Remediation Therapy on neuropsychological function, symptoms of eating disorders and general mental health, quality of life and motor activity in women with both eating disorders (transdiagnostic) and these specific cognitive difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Being in in-patient-, day- or out-patient treatment for an eating disorder (anorexia nervosa, bulimia nervosa, binge eating disorder or OSFED)
* Displaying cognitive difficulties (score ≤ -1 standard deviation) on:

  1. the Inhibit, Shift, Plan/ Organize and/ or Global Executive Composite indexes of the self-report measure the BRIEF-A (reversed)
  2. the Total errors, Perseverative Responses, Perseverative Errors and/ or Learning to learn from the Wisconsin Card Sorting Test (WCST) and/ or on the Rey Complex Figure Test (RCFT) Copy condition or Q-score and/ or on condition 3 and 4 on the Color-word Interference Test from (D-KEFS)
* Being able to understand and speak Norwegian
* Be willing to provide written informed consent
* Accepting random allocation to the two arms of the study

Exclusion Criteria:

* A history of congenital or acquired brain injury (except concussions)
* Active substance abuse
* Psychosis
* Intelligence quotient (IQ) less than 70

Ages: 16 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
BRIEF-A | 6 month follow-up
  Executive function according to the self-report questionnaire the Behaviour Rating Inventory of Executive Function, Adult (BRIEF-A). This questionnaire consist of 75 items on which the patient's symptoms are rated on a 3-point Likert scale. The questionnaire provides a Global Executive Composite score (range 75-225) and two index scores: the Behavioral Regulation Index (range 30-90) and the Metacognitive Index (range 40-120) in addition to nine subscales: Inhibit (range 8-24), Shift (range 6-18), Emotional control (range 10-30), Self-monitor (range 6-18), Initiate (range 8-24), Working memory (range 8-24), Plan/organize (range 10-30), Task monitor (range 6-18) and Organization of materials (range 8-24). Higher scores indicate more executive difficulties.
EDI-3 | 6 month follow-up
  Eating disorder- and general psychological symptoms according to the Eating Disorder Inventory, 3rd version (EDI-3). EDI-3 consist of 91 items rated on a 6 point Likert scale. The items are organized in to 12 primary scales: Drive For Thinness (range 0-28), Bulimia (range 0 -32), Body Dissatisfaction (range 0-40), Low Self-Esteem (range 0-24), Personal Alienation (range 0-28), Interpersonal Insecurity (range 0-28), Interpersonal Alienation (range 0-28), Interoceptive Deficits (range 0-36), Impulse Disregulation (range 0- 32), Perfectionism (range 0-24), Asceticism (range 0-28) and Maturity Fears (range 0-32). In addition, the EDI-3 also provides 6 composites: Eating Concerns Composite (range 0-100), Ineffectiveness (range 0-48), Interpersonal Problems (range 0- 52), Affective Problems (range 0-62), Overcontrol (range 0-52) and Global Psychological Maladjustment (range 0-252). Higher scores indicates more severe problems.
EDE-Q | 6 month follow-up
  Eating disorder behaviors (binge eating and inappropriate weight compensatory behaviors) and attitudinal features of eating disorders over the previous 28 days is measured by the Eating Disorder Examination (EDE-Q), v. 16.0. The EDE-Q includes 22-attitudinal items that are each rated using seven-point forced-choice format. The items are grouped into four clinically-derived subscales each consisting of five to eight items: Dietary restraint, Eating concern, Weight concern, and Shape concern. The score of each subscale is calculated as the average of item scores within the subscale and yields a range of 0-6. The global score is calculated as the average of the four subscale scores (range 0-6). Higher scores indicates greater pathology.
EDFLIX | 6 month follow-up
  Mental flexibility is measured according to the self-report questionnaire the Eating Disorder Flexibility Index (EDFLIX). This questionnaire consist of 36 items scored on a 6-point Likert scale. The questionnaire provides a total score (range 36-216) and three index scores: EDFLIX-GF (General Flexibility; range 17-102), EDFLIX-FoEx (Food and Exercise Flexibility; range 13-78) and EDFLIX-WeSh (Weight and Shape Flexibility; range 6-36). Higher scores indicate more flexibility.
WCST | 6 month follow-up
  Mental flexibility as measured by the Wisconsin Card Sorting Test (WCST)
RCFT | 6 month follow-up
  Central coherence as measured by the Rey Complex Figure Test (RCFT)
CWIT | 6 month follow-up
  Inhibition as measured by the Color-Word Interference Test (CWIT)

SECONDARY OUTCOMES:
SF-36v2 | 6 month follow-up
  Health related quality of life (HRQOL) was measured according to the Medical Outcomes Short-Form 36-Item Health Survey (SF-36v2). This questionnaire consist of 36 items on which the patient's responses are rated on a 3-point (item 3), 5-point (item 1, 2, 4, 5, 6, 8, 9, 10 and 11) or 6-point scale (item 7). The items are organized into eight domains: Physical Functioning (PF; 10 items), Role- Physical (4 items), Bodily Pain (BP; 2 items), General Health (GH; 5 items), Vitality (VT; 4 items), Social Functioning (SF; 2 items), Role- Emotional (3 items), and Mental Health (5 items). Furthermore, two summary measures can be calculated: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Transformed scores are calculated and yields a range of 0-100 for each domain- or summary measure. Higher scores indicate better HRQOL.
TMT | Post-intervention (12 weeks after baseline assessment), 6 month follow-up
  Performance on the Trail Making Test (TMT)
IGT | Post-intervention (12 weeks after baseline assessment), 6 month follow-up
  Performance on the Iowa Gambling Task (IGT)
Tower Test | Post-intervention (12 weeks after baseline assessment), 6 month follow-up
  Performance on the Tower Test
CCPT-3 | Post-intervention (12 weeks after baseline assessment), 6 month follow-up
  Performance on Conner's Continuous Performance Test- 3rd Edition (CCPT-3)
BDI-II | Post-intervention (12 weeks after baseline assessment), 6 month follow-up, 2 year follow-up
  Symptoms of depression according to the self-report questionnaire the Beck Depression Inventory- Second edition (BDI-II). This questionnaire consist of 21 items scored on a 4-point Likert scale (range 0- 63). Higher scores indicate more depression
BAI | Post-intervention (12 weeks after baseline assessment), 6 month follow-up, 2 year follow-up12 weeks (post-treatment)
  Symptoms of anxiety according to the self-report questionnaire the Beck Anxiety Inventory (BAI). This questionnaire consist of 21 items scored on a 4-point Likert scale (range 0- 63). Higher scores indicate more anxiety.
MCQ-30 | Post-intervention (12 weeks after baseline assessment), 6 month follow-up, 2 year follow-up
  Metacognitions as measured according to the Metacognitions questionnaire (MCQ-30). This questionnaire consist of 30 items scored on a 4-point Likert scale. The questionnaire provides a total score (range 30- 120) and 5 subscales: Positive beliefs about worry (range 6-24); Negative beliefs about worry concerning uncontrollability and danger (range 6-24), Cognitive confidence (range 6-24); Need to control thoughts (range 6-24) and Cognitive self-consciousness (range 6-24). Higher scores indicate more dysfunctional metacognitions.
Actigraphy | 6 months
  Actigraphy outcome measures from software
BRIEF-A | Post-intervention (12 weeks after baseline assessment), 2 year follow-up
  Executive function according to the self-report questionnaire the Behaviour Rating Inventory of Executive Function, Adult (BRIEF-A). This questionnaire consist of 75 items on which the patient's symptoms are rated on a 3-point Likert scale. The questionnaire provides a Global Executive Composite score (range 75-225) and two index scores: the Behavioral Regulation Index (range 30-90) and the Metacognitive Index (range 40-120) in addition to nine subscales: Inhibit (range 8-24), Shift (range 6-18), Emotional control (range 10-30), Self-monitor (range 6-18), Initiate (range 8-24), Working memory (range 8-24), Plan/organize (range 10-30), Task monitor (range 6-18) and Organization of materials (range 8-24). Higher scores indicate more executive difficulties.
EDI-3 | Post-intervention (12 weeks after baseline assessment), 2 year follow-up
  Eating disorder- and general psychological symptoms according to the Eating Disorder Inventory, 3rd version (EDI-3). EDI-3 consist of 91 items rated on a 6 point Likert scale. The items are organized in to 12 primary scales: Drive For Thinness (range 0-28), Bulimia (range 0 -32), Body Dissatisfaction (range 0-40), Low Self-Esteem (range 0-24), Personal Alienation (range 0-28), Interpersonal Insecurity (range 0-28), Interpersonal Alienation (range 0-28), Interoceptive Deficits (range 0-36), Impulse Disregulation (range 0- 32), Perfectionism (range 0-24), Asceticism (range 0-28) and Maturity Fears (range 0-32). In addition, the EDI-3 also provides 6 composites: Eating Concerns Composite (range 0-100), Ineffectiveness (range 0-48), Interpersonal Problems (range 0- 52), Affective Problems (range 0-62), Overcontrol (range 0-52) and Global Psychological Maladjustment (range 0-252). Higher scores indicates more severe problems.
EDE-Q | Post-intervention (12 weeks after baseline assessment), 2 year follow-up
  Eating disorder behaviors (binge eating and inappropriate weight compensatory behaviors) and attitudinal features of eating disorders over the previous 28 days is measured by the Eating Disorder Examination (EDE-Q), v. 16.0. The EDE-Q includes 22-attitudinal items that are each rated using seven-point forced-choice format. The items are grouped into four clinically-derived subscales each consisting of five to eight items: Dietary restraint, Eating concern, Weight concern, and Shape concern. The score of each subscale is calculated as the average of item scores within the subscale and yields a range of 0-6. The global score is calculated as the average of the four subscale scores (range 0-6). Higher scores indicates greater pathology.
EDFLIX | Post-intervention (12 weeks after baseline assessment), 2 year follow-up
  Mental flexibility is measured according to the self-report questionnaire the Eating Disorder Flexibility Index (EDFLIX). This questionnaire consist of 36 items scored on a 6-point Likert scale. The questionnaire provides a total score (range 36-216) and three index scores: EDFLIX-GF (General Flexibility; range 17-102), EDFLIX-FoEx (Food and Exercise Flexibility; range 13-78) and EDFLIX-WeSh (Weight and Shape Flexibility; range 6-36). Higher scores indicate more flexibility.
WCST | Post-intervention (12 weeks after baseline assessment), 2 year follow-up
  Mental flexibility as measured by the Wisconsin Card Sorting Test (WCST)
RCFT | Post-intervention (12 weeks after baseline assessment), 2 year follow-up
  Central coherence as measured by the Rey Complex Figure Test (RCFT)
CWIT | Post-intervention (12 weeks after baseline assessment), 2 year follow-up
  Inhibition as measured by the Color-Word Interference Test (CWIT)

CONTACTS AND LOCATIONS:
Overall Officials: Ute Gabriel, PhD, Study Director — Norwegian University of Science and Technology
Locations (3):
- Norway (3):
  - Levanger Hospital, Nord-Trøndelag Hospital Trust, Levanger, N-T
  - Department of Psychology, Norwegian University of Science and Technology, Trondheim
  - St Olavs Hospital HF, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thorsrud T, Thorsen L, Hjemdal O, Dahlgren CL, Micali N, Weider S. Neuropsychological Profiles in Patients With Restrictive or Binge/Purge Subtype Eating Disorders: A Continuum Approach. Eur Eat Disord Rev. 2026 Jan;34(1):178-190. doi: 10.1002/erv.70019. Epub 2025 Jul 29. PMID 40734305
- [Derived] Thorsrud T, Bang MA, Dahlgren CL, Nordfjaern T, Weider S. Cognitive remediation therapy for patients with eating disorders: a qualitative study. J Eat Disord. 2024 Sep 13;12(1):142. doi: 10.1186/s40337-024-01101-0. PMID 39272210